CLINICAL TRIAL: NCT06696183
Title: Sequential Gilteritinib in Combination With Venetoclax and Azacitidine for Patients With Newly Diagnosed Acute Myeloid Leukemia (AML) and FLT3 Mutations Ineligible for Intensive Treatment
Brief Title: Gilteritinib in Combination With Venetoclax and Azacitidine for AML Patients With FLT3 Mutations Ineligible for Intensive Treatment
Acronym: SEQUENCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-SEQUNC-081
Record Dates: First submitted 2024-11-07; First posted 2024-11-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: AML - Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): GILT d1-d28 VEN d1-d7 AZA d1-d7
  Interventions: Drug: Gilteritinib (GILT); Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)
- Cohort 2 (Experimental): GILT d8-d28 VEN d1-d7 AZA d1-d7
  Interventions: Drug: Gilteritinib (GILT); Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)
- Cohort 3 (Experimental): GILT d1-d28 VEN d1-d14 AZA d1-d7
  Interventions: Drug: Gilteritinib (GILT); Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)
- Cohort 4 (Experimental): GILT d8-d28 VEN d1-d14 AZA d1-d7
  Interventions: Drug: Gilteritinib (GILT); Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)

INTERVENTIONS:
Drug: Gilteritinib (GILT) — 80 mg
Drug: Venetoclax (VEN) — 400 mg
Drug: Azacitidine (AZA) — 75 mg/m²

SUMMARY:
Explore the best tolerable and efficacious dose of Gilteritinib when combined with standard treatment with Venetoclax and Azacitidine in AML patients with FLT3 mutations which are ineligible for intensive chemotherapy

ELIGIBILITY:
Main Inclusion Criteria:

* Newly diagnosed AML (according to WHO 2022 or ICC 2022 criteria) with a minimum BM blast count of >=20%, excluding APL
* FLT3 mutation at initial diagnosis
* Ineligibility of standard induction chemotherapy
* Pre-treatment with approved combination of Venetoclax + Azacitidine (one cycle only)

Main Exclusion Criteria:

* R/R AML
* Previous treatment for AML (except HU and/or one cycle VEN+AZA according to SOC)
* Previous treatment with Gilteritinib
* Known active CNS involvement
* QTcF >450 ms or long QT Syndrome at screening
* Treatment with concomitant strong CYP3A inducers or St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Ratio of dose delivered/dose planned | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided